CLINICAL TRIAL: NCT02665715
Title: Can Postprandial Reactive Hypoglycaemia be Reduced in Patients After Roux-en-Y Gastric Bypass With a Low Carbohydrate Diet?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amirsalar Samkani (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Sponsor-Investigator, Amirsalar Samkani, PhD-Student, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DK-REAKTIV-15
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Bariatric Surgery (Gastric Bypass)
Keywords: Reactive hypoglycemia; Hyperinsulinaemia; Diet; Glucagon-like Peptide-1; Glucagon; Peptide YY; Ghrelin
MeSH Terms: conditions — Hypoglycemia; Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low carbohydrate/Standard carbohydrate (Experimental): 10 Roux-en-Y gastric bypass operated subjects are tested two days with mixed-meal tests. Each studytest day consist of both breakfast and lunch.
  Interventions: Other: Low carbohydrate meals; Other: Standard carbohydrate meals
- Standard carbohydrate/Low carbohydrate (Experimental): 10 Roux-en-Y gastric bypass operated subjects are tested two days with mixed-meal tests. Each studytest day consist of both breakfast and lunch.
  Interventions: Other: Low carbohydrate meals; Other: Standard carbohydrate meals

INTERVENTIONS:
Other: Low carbohydrate meals — Meal macronutritional energy composition: Carbohydrate 30% Protein 30% Fat 40%
Other: Standard carbohydrate meals — Meal macronutritional energy composition: Carbohydrate 55% Protein 15% Fat 30%

SUMMARY:
Roux-en-Y gastric bypass (RYGB) accelerates nutrient delivery to the small intestine causing higher peak blood glucose concentration early after meal intake. In the late postprandial period (1 1⁄2-2 h) nadir blood glucose level is lower compared with before operation. In some patients, overt postprandial hypoglycaemia develops, and is typically reported as a complication 1-5 years postoperatively, when maximal weight loss has been obtained. The pathophysiology of postprandial hypoglycaemia involves inappropriate hyper-secretion of insulin associated with exaggerated secretion of the gut hormone glucagon-like peptide-1 (GLP-1) leading to a mismatch between glucose absorption rate, insulin secretion and whole body glucose disposal. We hypothesize that lowering carbohydrate content of meals reduces postprandial glucose excursions whereby GLP-1 and insulin secretion is reduced and reactive hypoglycemia prevented.

ELIGIBILITY:
Inclusion Criteria:

* RYGB operated patients more than 12 month after operation
* Stable in weight for at least 3 months (+/- 3 kg)
* Plasma glucose below 3.4 mmol/L after screening with test meal (Fresubin drink) or with continuous glucose monitoring

Exclusion Criteria:

* Fasting plasma glucose concentration > 7mmol/L
* Critical illness
* Hgb < 6.5 mM
* Pregnancy or breastfeeding

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Nadir plasma glucose | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.

SECONDARY OUTCOMES:
Peak plasma glucose | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.
Time to nadir glucose | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.
Time to peak glucose | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.
Postprandial incremental glucose area | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.
Postprandial decremental glucose area | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.
Postprandial incremental insulin area | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.
Postprandial incremental GLP-1 area | 0-240 min, 240-480 min
  Between low carbohydrate meal and standard meal.
Time below basline glucose concentrations | 0-480 min
  Between low carbohydrate meal and standard meal.
Glycemic excursions | 0-480 min
  Between low carbohydrate meal and standard meal.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine Bojsen-Moller, MD, Postdoc, Principal Investigator — Hvidovre University Hospital; Sten Madsbad, MD, Prof, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Endocrinology Research Center, Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Kandel D, Bojsen-Moller KN, Svane MS, Samkani A, Astrup A, Holst JJ, Madsbad S, Krarup T. Mechanisms of action of a carbohydrate-reduced, high-protein diet in reducing the risk of postprandial hypoglycemia after Roux-en-Y gastric bypass surgery. Am J Clin Nutr. 2019 Aug 1;110(2):296-304. doi: 10.1093/ajcn/nqy310. PMID 30624666